CLINICAL TRIAL: NCT04067726
Title: Randomized Clinical Trial of RANKL Inhibition With Denosumab on Mammographic Density in Premenopausal Women With Dense Breasts (TRIDENT)
Brief Title: RANKL Inhibition and Mammographic Breast Density
Acronym: TRIDENT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201907039
Record Dates: First submitted 2019-08-16; First posted 2019-08-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Dense Breasts
Keywords: Mammographic density; Breast cancer; RANKL; Denosumab; Prevention; Premenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab; Calcium; Cholecalciferol; Biopsy, Large-Core Needle; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Stratified permuted block randomized design will be used to generate the randomization table where permuted block randomization will be used for each stratum by age, with a varying block size of 4 and 6.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab (Experimental): * Subcutaneous injection of denosumab at a dose of 60 mg at two time points: baseline and 6 months
  * Participants will also be instructed to take calcium and vitamin D supplements daily for 12 months between baseline examination and 12-month mammographic breast density examination.
  * Mammographic breast density will be assessed at three time points in all participants: baseline, 12 months, and 24 months. A 36-month optional assessment may also occur.
  * Biopsies and blood draws will occur for research purposes at baseline and 12 months.
  Interventions: Drug: Denosumab; Drug: Calcium; Drug: Vitamin D3; Procedure: Core needle biopsy; Procedure: Blood draw
- Placebo (Placebo Comparator): * Subcutaneous injection of the placebo at a dose of 60 mg at two time points: baseline and 6 months
  * Participants will also be instructed to take calcium and vitamin D supplements daily for 12 months between baseline examination and 12 month mammographic breast density examination
  * Mammographic breast density will be assessed at three time points in all participants: baseline, 12 months, and 24 months. A 36 month optional assessment may also occur.
  * Biopsies and blood draws will occur for research purposes at baseline and 12 months.
  Interventions: Drug: Placebo; Drug: Calcium; Drug: Vitamin D3; Procedure: Core needle biopsy; Procedure: Blood draw

INTERVENTIONS:
Drug: Denosumab — Denosumab is commercially available and will be provided at no cost to participants.
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo — Placebo will be made available as 1 mL sterile, non-pyrogenic water solution in a single-use prefilled syringe.
  Arms: Placebo
Drug: Calcium — -Participants will be instructed to take calcium (at least 500 mg) daily for 12 months between baseline examination and 12- month mammographic breast density examination.
Drug: Vitamin D3 — Participants will be instructed to take vitamin D3 (at least 400 IU) supplements daily for 12 months between baseline examination and 12- month mammographic breast density examination.
Procedure: Core needle biopsy — Baseline and 12 months
Procedure: Blood draw — Baseline and 12 months

SUMMARY:
Data supporting a role for RANKL signaling in mammographic density and breast cancer development has begun to emerge, but clinical trial data providing definitive evidence that would allow the adoption of RANKL inhibition in primary breast cancer prevention are not yet available. The hypothesis is that RANKL inhibition with denosumab will decrease mammographic density in high-risk premenopausal women with dense breasts. To address this, the investigators have developed this clinical trial to quantify the impact of RANKL inhibition on mammographic density in high-risk premenopausal women with dense breasts and to determine the effect of RANKL inhibition on markers of proliferation and biomarkers of breast cancer risk. Successful demonstration that RANKL inhibition reduces mammographic density could open up additional approaches to primary breast cancer prevention in high-risk premenopausal women, who do not have dominant genetic predisposition.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Premenopausal (when menopausal status is uncertain, the investigators will measure follicle-stimulating hormone and estradiol to ascertain that a partcipant is premenopausal)
* At least 40 years of age.
* Dense breasts on routine mammogram (BI-RADS Category C and D)
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* History of breast or any other invasive cancer except for DCIS (ductal carcinoma in situ) who received only lumpectomy, LCIS (lobular carcinoma in situ), atypical hyperplasia, non-melanoma skin cancer, carcinoma in situ of the cervix.
* Current use of tamoxifen, aromatase inhibitors, or bisphosphonates, or RANKL inhibitors
* Concurrent participation in another cancer chemoprevention trial (unless no longer receiving the intervention).
* Pregnant, lactating, or planning to get pregnant while the trial is ongoing.
* Recent history of invasive dental procedure (e.g. tooth extraction, dental implant, oral surgery).
* Unhealed and/or planned dental/oral surgery.
* History of osteonecrosis/osteomyelitis of the jaw.
* History of osteoporosis or severe osteopenia.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in mammographic breast density between the two arms as measured by volumetric percent density | From baseline to 12 months
  -The investigators will use volumetric percent density (VPD) as the primary mammographic breast density measure.

SECONDARY OUTCOMES:
Change in mammographic breast density between the two arms as measured by volumetric percent density | From baseline to 24 months
Change in mammographic breast density between the two arms as measured by volumetric percent density | From 12 months to 24 months
Change in expression gene related to RANK in breast tissue compared between the two arms | Baseline and 12 months
Change in expression gene related to progesterone in breast tissue compared between the two arms | Baseline and 12 months
Change in expression gene related to metabolics in breast tissue compared between the two arms | Baseline and 12 months
Change in expression gene related to immune in breast tissue compared between the two arms | Baseline and 12 months
Change in expression gene related to inflammatory in breast tissue compared between the two arms | Baseline and 12 months
Change in expression of markers of breast epithelial and stromal proliferation compared between the two arms | Baseline and 12 months
Change in breast metabolome compared between the two arms | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adetunji T Toriola, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data used in generating tables and figures in published manuscripts.
Time Frame: IPD will be shared beginning 12 months, and ending 24 months following article publication.
Access Criteria: IPD will be shared with investigators who propose a methodologically sound proposal. These proposals should have been reviewed and approved by independent review committees, including institutional review boards. Proposals should be directed to the Principal Investigator, who will review the request with other co-Investigators. Proposals may also be subject to further review by the Protocol Review Monitoring Committee and Institutional Review Board at Principal Investigator's institution. Requestors will need to sign an institutional data access agreement to gain access to the data.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT04067726/ICF_000.pdf